CLINICAL TRIAL: NCT02517060
Title: Neural Mechanisms of Tactile Priming on Social Perceptions - Pilot Study
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Medical School Berlin (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Other Study IDs: SozPrime
Record Dates: First submitted 2015-07-10; First posted 2015-08-06 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Social perceptions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy participants: Male or female healthy participants

SUMMARY:
The investigators measure brain responses of healthy participants while they perform evaluation tasks inside the fMRI. For each task the participants were primed with tactile stimuli. Results should demonstrate engagement of sensorimotor brain regions after priming, hence confirming embodiment theories.

DETAILED DESCRIPTION:
Brain responses of healthy participants were recorded with functional magnetic resonance imaging (fMRI). While being scanned participants were asked to recommend punishments similar to judges or juries for perpetrators across different scenarios. In addition, participants were primed before reading the scenario by using different materials. Based on recent theories about "embodied cognition" and extralegal factors investigators hypothesize that those primes may influence the harshness of punishments recommended by the participants. If those processes engage sensorimotor cortices, the results would strongly support theories of embodied cognition.

The results would help the investigators to understand the neural correlates of priming processes. These unconscious complex processes of perception may be important for hospital patients. Thus, beneficial haptic experiences during the hospital stay may contribute to successful recovery.

ELIGIBILITY:
Inclusion Criteria:

* male or female healthy participants
* age 18 - 40 years

Exclusion Criteria:

* cardiac pacemaker
* metallic implants
* ferromagnetic parts in / at the body
* tatoos
* vessel surgery
* tinnitus
* epilepsia
* claustrophobia
* pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult male and female subjects
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Sensorimotor brain activation | The participantes will be followed up for the duration of fMRI-scan, an exspected average of 1 hour
  The primary objective of this study is to examine neural correlates for embodied cognitions. We use an fMRI-approach to test if healthy participants are prone to non-conscious tactile priming effects during evaluation processes. Investigators measure the outcome by examining BOLD Response in the sensorimotor cortices (Maximum Peak in Primary somatosensory Cortex, SI). BOLD Responses will be analyzed using the Software SPM 8.

SECONDARY OUTCOMES:
Systematic changes for evaluation processes | The participants will be followed up for the duration of fMRI-scan, an exspected average of 1 hour
  1. We examine if tactile priming leads to systematic behavioral changes for evaluation processes. During the fMRI participants were asked to read scenarios and subsequently perform evaluation processes on a likert scale 0 to 5 (0 = mild punishment; 5 = hard punishment) .

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (3):
- Germany (3):
  - Department of Psychiatry und Psychotherapy, CCM, Charité - University Medicine Berlin, Berlin, State of Berlin
  - Medical School Berlin, Berlin, State of Berlin
  - Department of Anesthesiology and Intensvie Care Medicine CVK/CCM, Charité - University Medicine Berlin, Berlin, State of Berlin